CLINICAL TRIAL: NCT00293904
Title: Safety, Immunogenicity and Clinical Efficacy of an Allergen Vaccine (CYT005-AllQbG10) in Subjects With Seasonal Rhinoconjunctivitis Due to Grass-Pollen Allergy
Brief Title: Safety and Efficacy of an Allergen Vaccine in Grass-Pollen Allergy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYT005-AllQbG10 02
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Hypersensitivity
Keywords: Allergy; Grass Pollen; Systemic Immunotherapy
MeSH Terms: conditions — Hypersensitivity

INTERVENTIONS:
Biological: CYT005-AllQbG10

SUMMARY:
The purpose of this study is to evaluate whether the use of a specific immunomodulatory principle (QbG10) together with conventional grass pollen allergen leads to a more rapid and more pronounced decrease of sensitivity against pollen than with the grass pollen allergen alone

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* Mild to moderate seasonal allergic rhinoconjunctivitis due to sensitization against grass pollen as evident from history (≥ 2 years), and positive nasal provocation test (NPT) and positive skin prick test (SPT, wheal ≥ 3mm larger than diluent) to grass pollen extract
* Female participants must meet one of the following criteria:

No reproductive potential due to menopause (one year without menses, in case of doubts serum FSH will be determined and must be >40 U/mL), hysterectomy, bilateral oophorectomy, or tubal ligation. Patient agrees to consistently practice an effective and accepted method of contraception throughout the duration of the study and for 1 additional months after the last immunization (hormone-based, or intrauterine device, or double barrier contraception, i.e. condom + diaphragm, condom or diaphragm + spermicidal gel or foam)

* Written informed consent
* Patient is willing and able to comply with all trial requirements

Exclusion Criteria:

* Additional allergies (seasonal or perennial) of which the symptoms overlap temporally with the screening and treatment period
* Contraindication to Allergen Preparation
* Contraindication for Nasal Provocation Test
* Contraindication for Skin Prick Test
* Actual significant obstructive pulmonary disorder (FEV1< 70%)
* Pharmacological treatment that could affect allergic sensitivity during the trial
* Presence or history of significant cardiovascular, renal, pulmonary, endocrine, autoimmune, neurological, and psychiatric disease as judged by the investigator
* Serum test positive for HIV, HBV, or HCV
* Current diagnosis or history of malignancy; presence of suspicious lymphadenopathy or splenomegaly on physical examination
* Pregnancy or lactation
* Blood donation within 30 days before enrolment
* History of abuse of alcohol or other recreational drugs
* Specific immunotherapy against pollen allergy within the last two years
* Intake of an investigational drug within three month before enrolment
* Intake of contraindicated medicaments for SIT as Betablockers, ACE/ATII Inhibitors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2006-02; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Nasal Provocation Tests

SECONDARY OUTCOMES:
Allergy and Medication Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Senti, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital of Zürich, Zurich, Canton of Zurich, Switzerland